CLINICAL TRIAL: NCT03485482
Title: Pharmacokinetic Drug-Drug Interaction Between Bisoprolol and Ivabradine in Healthy Volunteers: An Open-Label, Randomized, Crossover Clinical Study
Brief Title: Pharmacokinetic Drug-Drug Interaction Between Bisoprolol and Ivabradine in Healthy Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Mahmoud Shaheen, Associate Professor, Faculty of pharmacy, Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PHCL36
Record Dates: First submitted 2018-03-24; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Cardiovascular Diseases
Keywords: Pharmacokinetic drug interaction; ivabtadine; bisoprolol
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Bisoprolol; Ivabradine

STUDY DESIGN:
Intervention Model Description: open label, randomized, single-dose, three-period, crossover design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Ivabradine (Experimental): six healthy volunteers will administer Ivabradin tablet only once single 10 mg oral dose
  Interventions: Drug: Ivabradine
- Group Bisoprolol (Experimental): six healthy volunteers will administer bisoprolol tablet only once single oral dose of 5mg
  Interventions: Drug: Bisoprolol
- Group combination (Experimental): six healthy volunteers will administer only once a combination of a single dose of ivabradine 10 mg and bisoprolol 5 mg
  Interventions: Drug: combination of Ivabradine and bisoprolol

INTERVENTIONS:
Drug: Bisoprolol — bisoprolo 5 mg tablets
  Other Names: Concor
  Arms: Group Bisoprolol
Drug: Ivabradine — Ivabradine 10 mg tablet
  Other Names: Procorloan
  Arms: Group Ivabradine
Drug: combination of Ivabradine and bisoprolol — combination of 10 mg ivabradine and 5 mg bisoprolol
  Other Names: concor plus procorolan
  Arms: Group combination

SUMMARY:
The purpose of the study was to investigate the potential interaction between ivabradine and bisoprolol in healthy subjects.

DETAILED DESCRIPTION:
The aim of this study is to undergo a pharmacokinetic study to investigate the incidence of potential pharmacokinetic interaction between Ivabradine and Bisoprolol through the Assessment of the drug-drug interactions of Ivabradine and Bisoprolol by determination of pharmacokinetic parameters of both drugs administered alone and in combination. The pharmacokinetic parameters will include; The maximum plasma concentration (Cmax),the time to reach the peak concentration (tmax), area under the concentration-time curve (AUC0-t) and (AUC0-∞) during the treatment periods, the absorption and elimination rate constants (ka and kel), the half-life and mean residence time (MRT).

Study design A comparative randomized open-label three-period crossover study of ivabradine/ bisoprolol in male healthy human volunteers

Methodology

Eighteen healthy volunteer will be recruited in the study and will be divided into three groups each consisting of six volunteers as follows:

Period I:

* Group A: Six Volunteers will receive single 10 mg oral dose of ivabradin (Procoralan®, Les Laboratoires Servier Industrie-France).
* Group B: Six Volunteers will receive single oral dose of bisoprolol 5mg (Concor®).
* Group C: Six Volunteers will receive a single dose of ivabradine 10 mg and bisoprolol 5 mg

Period II:

* Group A: Six Volunteers will receive a single dose of ivabradine 10 mg and bisoprolol 5 mg
* Group B: Six Volunteers will receive single 10 mg oral dose of ivabradin.
* Group C: Six Volunteers will receive single oral dose of bisoprolol 5mg.

Period III:

* Group A: Six Volunteers will receive single oral dose of bisoprolol 5mg.
* Group B: Six Volunteers will receive a single dose of ivabradine 10 mg and bisoprolol 5 mg
* Group C: Six Volunteers will receive single 10 mg oral dose of ivabradin

All drug administration will be followed by 240 ml of water after at least 10 h fasting prior to administration. The three treatment periods will be separated by a one week washout period. Standardized meals will be served at 2, 5, and 10 h after drug dosing. All subjects should abstain from the consumption of fruit juices during the study period.

Subject Selection Criteria Eighteen adult male volunteers will be enrolled. Subjects should understand the procedures and are willing to participate and give their final written consent prior to the commencement of the study procedures.

ELIGIBILITY:
Inclusion Criteria:

Subjects should be healthy adult volunteers with age between (18-45 years) with normal body weight. Subjects should understand the procedures and are willing to participate and gave their final written consent prior to the commencement of the study procedures. The volunteers will be asked to provide a complete medical history, and complete a physical examination, laboratory tests [hematology, clinical chemistry, urinalysis, serology (including hepatitis B surface antigen, anti-hepatitis C virus and antihuman immunodeficiency virus antibody).

Exclusion Criteria:

1. Treatment with any known enzyme-inducing/inhibiting agents within 30 days prior to the start of the study and throughout the study.
2. Subjects who have taken any medication less than two weeks of the trials starting date.
3. Susceptibility to allergic reactions to study drugs.
4. Any prior surgery of the gastrointestinal tract that may interfere with drug absorption.
5. Gastrointestinal diseases.
6. Renal diseases.
7. Cardiovascular diseases.
8. Pancreatic disease including diabetes.
9. Hepatic diseases.
10. Hematological disease or pulmonary disease
11. Abnormal laboratory values.
12. Subjects who have donated blood or who have been involved in multiple dosing study requiring a large volume of blood (more than 500 ml) to be drawn within 6 weeks preceding the start of the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | 48 hours
  AUC0→∞
Pharmacokinetic parameters | 48 hours
  AUC0→t
Bioavailability parameters | 48 hours
  Cmax
Bioavailability parameters | 48 hours
  t max

CONTACTS AND LOCATIONS:
Overall Officials: Sara Shaheen, Ass. Prof, Principal Investigator — Faculty of pharamacy, Ain Shams University
Locations (1):
- Faculty of Pharmacy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No